CLINICAL TRIAL: NCT06216067
Title: Comparison of Operating Room Toric Placement Tools, CALLISTO Eye vs. Wavetec AnalyzOR (CORTCO)
Brief Title: Evaluate Performance of Callisto Eye vs. Wavetec AnalyzOR
Acronym: CORTCO
Status: Completed | Type: Observational
Sponsor: Chesapeake Eyecare and Laser Center, LLC (Other)
Collaborators: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Principal Investigator, Maria C. Scott, Dr. Maria C. Scott, MD, Chesapeake Eyecare and Laser Center, LLC
Other Study IDs: MCS12112021
Record Dates: First submitted 2023-12-20; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Cataract
Keywords: cataract; toric; cataract surgery; residual astigmatism
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Group 1 (Operating Room #1) CALLISTO eye: Group 1 (Operating Room #1) will have preoperative measurements with the IOL Master 700 and lens selection will be based on Veracity. The subjects in group 1 will have LenSx surgery and placement of the lens will be based on the CALLISTO eye.
  Interventions: Device: CALLISTO eye
- Group 2 (Operating Room #2) Wavetec AnalyzOR: Group 2 (Operating Room #2) will also have preoperative measurements with the IOL Master700, but lens selection will be based on the Wavetec AnalyzOR. The subjects in group 2 will have LenSx surgery and placement of the lens will be based on the Wavetec AnalyzOR.
  Interventions: Device: Wavetec AnalyzOR

INTERVENTIONS:
Device: CALLISTO eye — Cataract toric lens placement tool
  Groups: Group 1 (Operating Room #1) CALLISTO eye
Device: Wavetec AnalyzOR — Cataract toric lens placement tool
  Groups: Group 2 (Operating Room #2) Wavetec AnalyzOR

SUMMARY:
The goal of this clinical trial is to evaluate two separate operating room cataract measuring tools in predicting the residual astigmatism (prediction error) in patients with corneal astigmatism.

The main question it aims to answer is:

Show the refractive predictability comparing the use of Operating Room cataract toric lens placement tools against the standard manual technique.

Participants will be implanted with the TECNIS Toric II IOL Lens Model ZCU; the second eye, if applicable, is to be implanted within 45 days of the first-eye surgery.

Researchers will compare two Operating Room cataract lens placement tools: the Zeiss CALLISTO vs. the Wavetec AnalyzOR to determine refractive predictability.

DETAILED DESCRIPTION:
To evaluate two separate operating room cataract measuring tools in predicting the residual astigmatism (prediction error) in patients with corneal astigmatism (maximum allowable up to 3.0D) comparing the ZEISS CALLISTO eye and the Wavetec AnalyzOR at the one-month post-operative visit. Both surgery rooms will be using Veracity, IOL Master and Zeiss Opmi Lumera i Operating Room Microscopes. Operating Room #1 will be utilizing the ZEISS CALLISTO eye for axis alignment, along with Veracity and IOL Master for lens selection, and Operating Room #2 will be utilizing the Wavetec AnalyzOR for lens selection and axis alignment. Procedure times for the ZEISS CALLISTO eye and the Wavetec AnalyzOR will be obtained by using a start/stop watch, including phakic power calculation and toric positioning. In addition, the suction on (start of LenSx), treatment time of LenSx in seconds, suction off (end of LenSx), start time of primary incision, the beginning of Phaco, end of phaco, CDE (Combined Diffused Energy) total and the end time of procedure will all be documented. All times will be analyzed and compared between Operating Room #1 and Operating Room #2.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral cataract extraction with single piece hydrophobic acrylic posterior capsular intraocular lens correcting astigmatism.
* Clear intraocular media other than cataract.
* Willing and able to complete all required postoperative visits.
* Able to comprehend and sign a statement of informed consent in English.

Exclusion Criteria:

* Ocular disease or pathology that, in the opinion of the Investigator, will affect the post-operative visual acuity and manifest refraction.
* Prior intraocular or corneal refractive surgery, corneal transplant, or retinal detachment.

Ages: 55 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing unilateral or bilateral cataract extraction
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Diopters of Residual Cylinder | 1 Month postoperatively from implantation of intraocular lens
  Diopters of Residual Cylinder at Month 1 with an upper boundary and lower boundary of +0.50 D and - 0.50 D

SECONDARY OUTCOMES:
Accuracy of Residual Astigmatism (Predictive Error) | Month 1
  Residual Astigmatism of +/- 0.25 D or less, +/- 0.75 D or less, +/- 1.00 or less
Refractive predictability of the IOL (absolute difference between MRSE and target MRSE) | Month 1
  MRSE within 0.25, 0.50, 0.75, 1.00 of target
Uncorrected Distance Visual Acuities Achieved - Snellen | Month 1
  Achievement of UCDVA of 20/20, 20/25, 20/30, 20/40 or better
Procedure and Operating Room Time | Procedure time (up to 2 minutes)
  Suction on (start of LenSx), treatment time of LenSx in seconds, Suction off (end of LenSx)
Operating Room Time | Operating Room Time (up to 30 minutes)
  Start and end time of matching reference image to microscope image, start time-primary incision, beginning of Phaco, end of Phaco, CDE (Combined Diffused Energy) Total, Start and end time of phakic power calculation, start and end time of toric positioning, end time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Maria C. Scott, Principal Investigator — Chesapeake Eyecare and Laser Center, LLC
Locations (1):
- Chesapeake Eye Care and Laser Center, LLC, Annapolis, Maryland, United States

IPD SHARING:
Plan to Share IPD: No